CLINICAL TRIAL: NCT01506505
Title: A Randomised Controlled Cross-over Trial to Evaluate Evening Versus Morning Administration of a Cardiovascular Polypill
Brief Title: The Evening Versus Morning Polypill Utilization Study
Acronym: TEMPUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, dr.Frank L.J. Visseren, Clinical Professor, UMC Utrecht
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2011-001120-38
Record Dates: First submitted 2011-11-23; First posted 2012-01-10 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-08

CONDITIONS: Cardiovascular Disease; Cerebrovascular Disease; Peripheral Arterial Disease
Keywords: Cardiovascular prevention; Polypill; Combination therapy
MeSH Terms: conditions — Cardiovascular Diseases; Cerebrovascular Disorders; Peripheral Arterial Disease | interventions — Cardiovascular Agents; Aspirin; Simvastatin; Lisinopril

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Polypill in the morning (Experimental): Cardiovascular agents in a polypill used from 05.00-11.00 in the morning (acetylsalicylic acid 75 mg, simvastatin 40 mg, lisinopril 10 mg, hydrochlorothiazide 12,5 mg)
  Interventions: Drug: Cardiovascular Agents
- Polypill in the evening (Experimental): Cardiovascular agents in a polypill used from 18.00-00.00 in the evening (acetylsalicylic acid 75 mg, simvastatin 40 mg, lisinopril 10 mg, hydrochlorothiazide 12,5 mg)
  Interventions: Drug: Cardiovascular Agents
- Individual agents of the polypill) (Active Comparator): Cardiovascular agents in as acetylsalicylic acid 75 mg, lisinopril 10 mg, hydrochlorothiazide 12,5 mg used 05.00-11.00 in the morning.
  Simvastatin 40 mg used 18.00-00.00 in the evening.
  Interventions: Drug: Cardiovascular Agents

INTERVENTIONS:
Drug: Cardiovascular Agents — Acetylsalicylic acid 75mg, simvastatin 40mg, lisinopril 10mg, hydrochlorthiazide 12.5mg in individual agents or a combination pill
  Other Names: Acetylsalicylic acid 80 mg; Simvastatin 40 mg; Lisinopril 10 mg; Hydrochlorothiazide 12,5 mg

SUMMARY:
Background and rationale:

In clinical practice, antihypertensives are generally prescribed for use in the morning, whereas some statins are recommended for use in the evening. There is evidence that the reduction in LDL cholesterol achieved with some statins is superior when taken in the night, but it is unclear whether the additional reduction in LDL cholesterol(and the reported improvement in BP control when aspirin is taken in the evening) is offset by a reduction in adherence when taking medication in the evening. Current product labelling recommends night use for simvastatin and does not state a timing preference for aspirin or blood pressure lowering medicines. There is therefore uncertainty concerning the best timing of administration of the polypill. This uncertainty will be addressed by this trial.

Trial design:

Randomised, open label cross over trial (n=75) of the polypill in the morning compared with the evening administration compared with individual agent administration (acetylsalicylic acid and blood pressure lowering agents in the morning, and statin in the evening) in individuals at high risk of cardiovascular disease. Patients will be recruited to the RHP 2c (acetylsalicylic acid 75mg, simvastatin 40mg, lisinopril 10mg, hydrochlorthiazide 12.5mg), and will be randomly allocated to the sequence of time of administration.

DETAILED DESCRIPTION:
Background and rationale:

In clinical practice, antihypertensives are generally prescribed for use in the morning, whereas some statins are recommended for use in the evening. There is evidence that the reduction in LDL cholesterol achieved with some statins is superior when taken in the night, but it is unclear whether the additional reduction in LDL cholesterol(and the reported improvement in BP control when aspirin is taken in the evening) is offset by a reduction in adherence when taking medication in the evening. Current product labelling recommends night use for simvastatin and does not state a timing preference for aspirin or blood pressure lowering medicines. There is therefore uncertainty concerning the best timing of administration of the polypill. This uncertainty will be addressed by this trial.

Trial design:

Randomised, open label cross over trial (n=75) of the polypill in the morning compared with the evening administration compared with individual agent administration (acetylsalicylic acid and blood pressure lowering agents in the morning, and statin in the evening) in individuals at high risk of cardiovascular disease. Patients will be recruited to the RHP 2c (acetylsalicylic acid 75mg, simvastatin 40mg, lisinopril 10mg, hydrochlorthiazide 12.5mg), and will be randomly allocated to the sequence of time of administration.

Aim:

To measure whether there is a difference in LDL cholesterol levels or the 24 hour ambulatory blood pressure in individuals at high risk of cardiovascular disease when the polypill is taken in the morning compared to the evening.

Randomisation and trial treatment:

Eligible individuals willing to participate in the trial will receive the polypill for a total of 18 weeks and be randomised to the sequence of 6 weeks morning, 6 weeks evening administration and 6 weeks administration of the individual agents. The polypill will be provided by the investigator at the Trial Centre. Participants will also receive information about smoking cessation (if applicable) and how to follow a healthy heart diet. They will be advised to increase physical activity and lose weight if needed.

Data collection and follow-up:

Participants will be followed-up for 20 weeks. Ambulatory blood pressure will be measured at baseline and week 6, week 12 and week 18. Fasting lipids will be measured at baseline, weeks 6, 12 and 18. Tolerability will be assessed at weeks 6, 12, 18 and 20 as will adverse events. Participant acceptability will be measured at the end of the treatment period.

Primary outcome:

Difference in LDL cholesterol and mean 24 hour ambulatory systolic BP.

ELIGIBILITY:
Inclusion Criteria:

* The participant is able to give informed consent.
* The trial Investigator considers that each of the polypill components are indicated at the doses in the Red Heart Pill
* Established atherothrombotic cardiovascular disease (CVD) or intermediate to high cardiovascular risk, defined as;

  * History of coronary heart disease (myocardial infarction, stable or unstable angina pectoris, or coronary revascularisation procedure), or
  * History of ischaemic cerebrovascular disease (ischaemic stroke or transient ischaemic attack), or
  * History of peripheral vascular disease (peripheral revascularisation procedure or amputation due to vascular disease or aortic reconstruction), or
  * For individuals without established cardiovascular disease, a calculated 5 year CVD risk of 5% or greater (calculated using the 1991 Anderson Framingham risk equation with adjustments as defined by the New Zealand Guidelines Group recommendations - (Appendix 1))

Exclusion Criteria:

* Contraindication to any of the components of the polypill (e.g. known intolerance to aspirin, statins, or ACE inhibitors; pregnancy or likely to become pregnant or breastfeeding women during the treatment period). Such contraindications are fully listed in the Investigator Brochures.
* The treating doctor considers that changing a participant's cardiovascular medications would put the participant at risk (e.g. symptomatic heart failure, high dose β-blocker required to manage angina or for rate control in atrial fibrillation, accelerated hypertension, severe renal insufficiency, a history of severe resistant hypertension).
* Other potential reasons for exclusion include:
* Known situation where medication regimen might be altered for a significant length of time, e.g. current acute cardiovascular event, planned coronary bypass graft operation.
* Unlikely to complete the trial (e.g. life-threatening condition other than cardiovascular disease) or adhere to the trial procedures or attend study visits (e.g. major psychiatric condition, dementia).
* Any reason, medical condition, ongoing medication or significant disability that would prevent the participant complying with trial consent, treatment and follow-up procedures or potentially jeopardise her / his medical care.
* Night shift workers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
LDL cholesterol (polypill evening vs polypill morning) | 24 weeks
  Differences between polypill in the evening (after 8 weeks of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) in:
  - Mean LDL cholesterol
Mean 24 hour ambulatory systolic BP (polypill evening vs morning) | 24 weeks
  Difference between the between polypill in the evening (after 8 weeks of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) in:
  - Mean 24 hour ambulatory systolic BP

SECONDARY OUTCOMES:
Differences in ambulatory BP parameters after a mean of 7 week of treatment (polypill evening vs. morning, polypill vs regular care) | 24 weeks
  Differences between polypill in the evening (after 8 weeks of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) and regular care (after 8 weeks of treatment with individual agents of the polypill) in:
  * Mean 24 hour ambulatory diastolic BP
  * Mean diurnal (awake) and nocturnal (asleep) systolic and diastolic BP.
  * Percentage of dipping of SBP.
Differences in tolerability (adverse event, cessation of treatment) | Every 6-8 weeks
  Difference between polypill in the evening (after 8 weeks of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) and regular care (after 8 weeks of treatment with individual agents of the polypill) in:
  * Patients' acceptability
  * Number of adverse events
  * Number of cessation of study treatment
Adherence (polypill evening vs. morning, polypill vs regular care) | 24 weeks
  Differences between polypill in the evening (after 8 of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) and regular care (after 8 weeks of treatment with individual agents of the polypill) in:
  * Patients' adherence measured with electronic medication registration lids (MEM spots, AARDEX group)
  * Patients' self reported adherence
Cholesterol fractions (polypill evening vs. morning, polypill vs regular care) | 24 weeks
  Differences between polypill in the evening (after 8 of evening treatment) and polypill in the morning (after 8 weeks of morning treatment) and regular care (after 8 weeks of treatment with individual agents of the polypill) in:
  * Mean total cholesterol.
  * Mean HDL cholesterol.
  * Mean triglycerides.
  * Mean total:HDL ratio

CONTACTS AND LOCATIONS:
Overall Officials: W. Spiering, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Lafeber M, Grobbee DE, Schrover IM, Thom S, Webster R, Rodgers A, Visseren FL, Bots ML, Spiering W. Comparison of a morning polypill, evening polypill and individual pills on LDL-cholesterol, ambulatory blood pressure and adherence in high-risk patients; a randomized crossover trial. Int J Cardiol. 2015 Feb 15;181:193-9. doi: 10.1016/j.ijcard.2014.11.176. Epub 2014 Dec 3. PMID 25528311
- [Derived] Lafeber M, Grobbee DE, Bots ML, Thom S, Webster R, Rodgers A, Visseren FL, Spiering W. The evening versus morning polypill utilization study: the TEMPUS rationale and design. Eur J Prev Cardiol. 2014 Apr;21(4):425-33. doi: 10.1177/2047487313476961. Epub 2013 Feb 4. PMID 23382539